CLINICAL TRIAL: NCT06794697
Title: Evaluation of Preoperative Anxiety Level Based on the Day of Admission for Cardiac Surgery
Acronym: ADMITY
Status: Recruiting | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC23_3034_ADMITY
Record Dates: First submitted 2025-01-06; First posted 2025-01-27 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Surgery
Keywords: preoperative anxiety; cardiac surgery; evaluation of anxiety; admission day; APAIS scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients admitted the day before their surgery (J-1): Patients admitted the day before their cardiac surgery (J-1) will be invited to complete the questionnaire in two stages : upon admission and just before leaving for the operating room
  Interventions: Other: Questionnaire including APAIS scale
- Patients admitted on the day of surgery (J-0): Patients admitted on the day of cardiac surgery (J-1) will be invited to complete the questionnaire in two stages : upon admission and just before leaving for the operating room
  Interventions: Other: Questionnaire including APAIS scale

INTERVENTIONS:
Other: Questionnaire including APAIS scale — Patients will complete a questionnaire in two stages : upon admission and just before leaving for the operating room

SUMMARY:
Prospective, observational, non-randomized study that evaluates the impact of the admission day (J-1 vs J-0) on preoperative anxiety in cardiac surgery patients.

DETAILED DESCRIPTION:
The goal of this study is to determine whether the admission day (J-1 or J-0) has a significant effect on preoperative anxiety using the APAIS (Amsterdam Preoperative Anxiety and Information) scale and to identify modifiable factors to improve patient care.

This study includes 400 patients divided into two groups : 200 patients admitted the day before their surgery (J-1) and 200 patients admitted on the day of surgery (J-0).

Patients admitted for cardiac surgery at the University Hospital of Rennes will be invited to participate after verification of the inclusion criteria. A nurse or surgeon will explain the objectives and procedures of the study and provide the patient with an information and non-opposition letter. If the patient agrees, they will be included in the study, and the non-opposition form will be recorded in their medical file.

Patients will complete the questionnaire in two stages : upon admission and just before leaving for the operating room. The estimated time to complete the questionnaire is approximately 15 minutes, with 10 minutes for the first part and 5 minutes for the second part.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years old
* Scheduled for cardiac surgery
* Have received written and oral information about the protocol
* Admitted to the cardiac and thoracic surgery units
* Not opposed to participating in the research.

Exclusion Criteria:

* Patient undergoing emergency cardiac surgery with no time for reflection
* Legal adults under legal protection (guardianship, curators, or legal protection)
* Pregnant or breastfeeding women, minors, individuals unable to express consent
* Patient on long-term anxiolytic treatment
* Patient with psychiatric disorders, cognitive impairments, or central neurological disorders.
* Patient already participating in an ongoing study in the department of Thoracic and Cardiovascular Surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cardiac pathology requiring cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Comparison of the level of anxiety before leaving for the operating room between patients arriving the day before the operation and those arriving on the day of the operation. | Day of scale completion
  Amsterdam Preoperative Anxiety and Information Scale (APAIS) - score 1 to 5 (1=not anxious at all ; 5=extremely anxious)

SECONDARY OUTCOMES:
Comparison of of the level of anxiety at admission and before leaving for the operating room between the 2 groups | Day of scale completion
  Amsterdam Preoperative Anxiety and Information Scale (APAIS) - score 1 to 5 (1=not anxious at all ; 5=extremely anxious)
Comparison of of the level of anxiety at admission and before leaving for the operating room between the 2 groups | Day of scale completion
  Answers to a questionnaire
Comparison of the level of preoperative anxiety before going to the operating room according to patient comfort parameters | Day of scale completion
  Amsterdam Preoperative Anxiety and Information Scale (APAIS) - score 1 to 5 (1=not anxious at all ; 5=extremely anxious)
Comparison of the level of preoperative anxiety before going to the operating room according to patient comfort parameters | Day of scale completion
  Answers to a questionnaire
Comparison of preoperative anxiety according to patient's understanding of the surgery and the type of surgical procedure | Day of scale completion
  Amsterdam Preoperative Anxiety and Information Scale (APAIS) - score 1 to 5 (1=not anxious at all ; 5=extremely anxious)
Comparison of preoperative anxiety according to patient's understanding of the surgery and the type of surgical procedure | Day of scale completion
  Answers to a questionnaire
Comparison of preoperative anxiety according to the surgical schedule | Day of scale completion
  Amsterdam Preoperative Anxiety and Information Scale (APAIS) - score 1 to 5 (1=not anxious at all ; 5=extremely anxious)
Comparison of preoperative anxiety according to the surgical schedule | Day of scale completion
  Answers to a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No